CLINICAL TRIAL: NCT02784938
Title: Randomized Clinical Trial Evaluating the Efficacy of the Peer-run Vocational Empowerment Photovoice (VEP) to Increase the Capacity of Individuals With Psychiatric Disabilities to Pursue Employment
Brief Title: Vocational Empowerment Photovoice (VEP)
Acronym: VEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); Thresholds Inc. (Industry); Pilgrim Psychiatric Center (Unknown)
Responsible Party: Principal Investigator, Zlatka Russinova, Research Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 90RT5029-01-00 R3
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Mental Illness
Keywords: Employment; Mental Illness; Photovoice
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vocational Empowerment Photovoice (VEP) (Experimental): The VEP program is a 10-week manualized, structured, peer-led intervention delivered in 2-hour group sessions. The VEP program integrates Photovoice methodology, Rehabilitation Readiness technology and elements of the Anti-Stigma Photovoice (ASP) curriculum previously developed and tested by the Boston University Center for Psychiatric Rehabilitation (BU CPR). VEP group sessions combine didactic information, Photovoice exercises, and group discussions to empower participants in pursuing employment services and opportunities, all refined with input from individuals with a lived experience.
  Interventions: Behavioral: Vocational Empowerment Photovoice (VEP)
- Wait-list Control (No Intervention): Services as usual

INTERVENTIONS:
Behavioral: Vocational Empowerment Photovoice (VEP) — The VEP program is a 10-week manualized, structured, peer-led intervention delivered in 2-hour group sessions. The VEP manual includes a Workbook for the clients and a corresponding Leader's Guide for the group peer-leaders. The VEP program integrates Photovoice methodology, Rehabilitation Readiness technology and elements of the Anti-Stigma Photovoice (ASP) curriculum previously developed and tested by the Boston University Center for Psychiatric Rehabilitation (BU CPR). VEP group sessions combine didactic information, Photovoice exercises, and group discussions to empower participants in pursuing employment services and opportunities, all refined with input from individuals with a lived experience.
  Arms: Vocational Empowerment Photovoice (VEP)

SUMMARY:
The purpose of this project is to evaluate a promising peer-run psycho-educational group intervention titled "Vocational Empowerment Photovoice (VEP)" that aims to empower individuals with the most disabling psychiatric disabilities to engage in vocational services and pursue employment through the enhancement of their vocational hope, sense of vocational identity, work motivation, work-related self-efficacy, and capacity to deal with psychiatric stigma and discrimination.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate a promising peer-run psycho-educational group intervention titled "Vocational Empowerment Photovoice (VEP)" that aims to empower individuals with the most disabling psychiatric disabilities to engage in vocational services and pursue employment through the enhancement of their vocational hope, sense of vocational identity, work motivation, work-related self-efficacy, and capacity to deal with psychiatric stigma and discrimination. The VEP program was designed and pilot tested with a small randomized study (n=51) as part of a National Institute of Disability and Rehabilitation Research (NIDRR) funded research and training center (RTC) on Improving the Employment Outcomes (2009-2014). VEP is a 10-week peer-run program enhanced with 3 group booster sessions and the availability of weekly individual support provided by the VEP peer-leaders in keeping with each participant's formulated vocational goals. The researchers propose to evaluate the effectiveness of the VEP intervention using a large multi-site randomized controlled trial (RCT) with a total of 160 individuals who are not engaged in vocational services or working, but express such interests. The RCT will be carried out at 2 different mental health agencies (Thresholds in Chicago, IL and Pilgrim Psychiatric Center in Long Island, NY) both of which provide supported employment services. Eighty individuals will be recruited at each of these two study sites and will be assessed at baseline and 4 post baseline follow-up points. The efficacy of the VEP intervention will be tested in regards to two types of outcomes: a) extrinsic (for example, engagement in employment services, job-seeking activities, or employment), and b) intrinsic (for example, enhanced vocational hope, sense of vocational identity, work motivation, work-related self-efficacy). The researchers propose a small qualitative sub-study to inform future implementation and scaling up of VEP based on its effectiveness. Upon completion of each wave of the RCT the researchers will conduct an approximately 90-minutes focus group with participants in the VEP program and individual interviews with the VEP peer leaders. At the conclusion of the RCT at each collaborating site, the researchers will conduct individual interviews with the VEP supervisor(s), research staff and agency senior manager(s) familiar with the study.

The study is currently approved for the Thresholds site and recruitment is under way at this site.

ELIGIBILITY:
Inclusion Criteria:

1. are 18 or older
2. have a DSM-IV diagnosis of serious mental illness, including dual diagnosis
3. are not working currently due to their mental illness
4. are not receiving or in a process of receiving employment services
5. are interested in learning about ways to pursue work in the future
6. are fluent in English.

Exclusion Criteria:

1. co-existing physical or developmental disabilities resulting in cognitive limitations
2. Inability to give full and knowing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Engagement in employment and employment services | Baseline to 12 months
  Measured by number of appointments with supported employment providers and days employed during each follow up period.
Work Hope | Baseline to 12 months
  Measured by the Work Hope Scale
Vocational Identity | Baseline to 12 months
  Measured by the Vocational Identity Scale
Work Motivation | Baseline to 12 months
  Measured by the Work Motivation Scale

SECONDARY OUTCOMES:
Belief in Work Capacity | Baseline to 12 months
  Measured by a single item scale
Internalized Stigma | Baseline to 12 months
  Measured by the Internalized Stigma of Mental Illness Scale
Empowerment | Baseline to 12 months
  Measured by Making Decisions Empowerment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Zlatka Russinova, Study Director — Boston University
Locations (3):
- United States (3):
  - Thresholds Inc., Chicago, Illinois
  - Baycove Human Services- Transitions of Boston, Dorchester, Massachusetts
  - Pilgrim Psychiatric Center, Brentwood, New York

IPD SHARING:
Plan to Share IPD: No